CLINICAL TRIAL: NCT03354481
Title: Automatization of Counting Procedures in Children With Dyscalculia
Acronym: PROCEDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0651; 2017-A03134-49 (Other: ANSM)
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dyscalculia
Keywords: Dyscalculia
MeSH Terms: conditions — Dyscalculia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral recording of arithmetic and associated information (Experimental): The experiment will contain several behavioral tasks in which solving time and correct answer will be recorded. The main one will be a computerized task on arithmetic facts. There will also be three additional tasks as described below.
  Interventions: Behavioral: Arithmetic facts solving

INTERVENTIONS:
Behavioral: Arithmetic facts solving — The experiment will contain several tasks. The main one will be a computerized task on arithmetic facts where participants will have to solve simple additions. There will also be three additional tasks: a processing speed task where the participant will have to tell the orientation of an arrow as fast as possible, a visuo-spatial task where the participant will have to reproduce a tapping block sequence and an arithmetic task where the participant will try to solve a maximum of operations in a limited time.

SUMMARY:
Researchers in numerical cognition usually think that the greatest and most common difficulty in children suffering from dyscalculia is retrieval of arithmetic facts from long-term memory. However, we have recently shown that retrieval might not be the optimum strategy in mental arithmetic. In fact, expert adults would rather solve simple problems such as 3 + 2 by automated and unconscious procedures. Therefore, we hypothesize that children with dyscalculia might not present deficit in retrieval but, instead, in counting procedure automatization. The aim of the current project is to test this challenging position. Through a longitudinal approach, we plan to precisely examine the behavior of children suffering from dyscalculia over a 3-year period. Children will be aged between 8 to 11 years at the beginning of the study and we will precisely observe the evolution of their solution times when they solve simple addition problems involving one-digit numbers. If children with dyscalculia still struggle with simple additions three years, their solution times plotted on the sum of the problems should still follow an exponential function. Indeed, if counting is not automated, difficulties necessarily increase with the progression on the number line or the verbal sequence, hence the exponential function. On the contrary, if counting procedures tend towards automatization, moves along a number line will progressively become as easy at the beginning of the line as at the end, hence the linear function. Importantly, a retrieval model would predict exactly the inverse pattern because, according to this model, the linear function, which is unanimously considered as the hallmark of counting procedures, should progressively be replaced by a non-linear function through practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 11 years old
* Having a dyscalculia as described in the DSM (Diagnostic and Statistical Manual) V

Exclusion Criteria:

* Presenting a global intellectual deficit

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Response times to solve an informatics task on simple arithmetic facts resolution | Inclusion
  Time between the apparition of the stimuli and the answer. The task contain only addition of one digit numbers
Response times to solve an informatics task on simple arithmetic facts resolution | 12 months
  Time between the apparition of the stimuli and the answer. The task contain only addition
Response times to solve an informatics task on simple arithmetic facts resolution | 24 months
  Time between the apparition of the stimuli and the answer. The task contain only addition

SECONDARY OUTCOMES:
Percentage of correct responses to solve the informatics task on simple arithmetic facts resolution | 0+ 12 + 24 months
Result of the digit span memory task | 0 month
Processing speed in an informatics task on arrow orientation | 0 month
Result of the Corsi block tapping test | 0 month
Result of the Tempo Test Rekenen | 0 month
  The Tempo Test Rekenen is used to evaluate arithmetical ability. It consists in solving several operations in a limited time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeanne Bagnoud, Romain Mathieu, Jasinta Dewi, Sandrine Masson, Sibylle Gonzalez-Monge, Zumrut Kasikci and Catherine Thevenot. An investigation of the possible causes of arithmetic difficulties in children with dyscalculia. L'Année psychologique 2021/3 Vol.121